CLINICAL TRIAL: NCT00789347
Title: Analysis of Cortical Excitability in Neuropathic Pain: an Electrophysiology Study.
Brief Title: Analysis of Cortical Excitability in Neuropathic Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sung-Tsang Hsieh/ MD. PHD., National Taiwan University, Department of Neurology
Other Study IDs: 200806061R
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-03

CONDITIONS: Neuropathic Pain; Cortical Excitability
Keywords: Neuropathic pain; Cortical excitability; Transcranial magnetic stimulation; Contact Heat evoked potential; peripheral nerve stimulation; neurotrophic factors
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Genomic polymorphism of neurotrophic factors.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Healthy volunteers
- 2: Patient with neuropathic pain
- 3: patients without neuropathic pain

SUMMARY:
The purpose of this study is to determine whether patients with neuropathic pain has abnormal excitability in somatosensory cortex and abnormal sensory-motor connections.

DETAILED DESCRIPTION:
There are several brain areas responsible for neuropathic pain reported in functional image studies, including primary sensory cortex, insula, and anterior cingulate gyrus. However, it is few informations about the functional status of these areas. Besides, the reason of the individual variability about the developement of neuropathic pain remains unknown. It is lack of satisfactory explanation about why some people developed neuropathic pain in certain diseased situation (for example, type 2 diabetes), while others do not.

We hypothesis that patients with neuropathic pain has abnormal cortical excitability and plasticity in certain brain area. Therefore developed neuropathic pain certain diseased condition while others not. Therefore, we will use multimodal electrophysiology tools,such as transcranial magnetic stimulation, peripheral nerve stimulation, and contact heat evoke potential to monitor the cortical excitability and plasticity non-invasively.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* patients with pain resulted from dysfunction of peripheral or central nervous system
* the disorders of peripheral nerves are diagnosed by nerve conduction study, quantitative sensory test, quantification of skin innervation or contact heat evoked potentials
* lesion of central nervous system should be confirmed by neuroimage.

Exclusion Criteria:

* previous history of epilepsy, seizure disorders or major head injury
* previous brain surgery or intracranial metalic implant
* implanted devices as cardiac pacemaker
* pregnant subjects
* patient with severe cardiac or pulmonary disease who potentially cannot tolerate stress

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic healthy volunteer
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2008-10; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Abnormal cortical excitability in motor-sensory cross-talk | non-applicable

SECONDARY OUTCOMES:
Genetic variability of neurotrophic factors between groups | non-applicable

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Kai Pan, M.D., Study Director — National Taiwan University Hospital, Department of Neurology; Chi-Chao Chao, M.D., Study Director — National Taiwan University Hospital, Department of Neurology; Sung-Tsang Hsieh, M.D. PhD, Principal Investigator — National Taiwan University Hospital, Department of Neurology
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan